CLINICAL TRIAL: NCT05889039
Title: Effects of Osteopathic Manipulative Treatment (OMT) and Bio Electro-Magnetic Regulation (BEMER) Therapy on Neck Pain in Adults
Brief Title: Effects of Osteopathic Manipulative Treatment and Bio Electro-Magnetic Regulation Therapy on Neck Pain in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lake Erie College of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Santiago Lorenzo, PhD, Professor of Physiology, Lake Erie College of Osteopathic Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 26-164
Record Dates: First submitted 2023-05-10; First posted 2023-06-05 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Neck Pain
Keywords: Neck Pain; Osteopathic Manipulative Treatment (OMT); BEMER
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- OMT + BEMER PLACEBO (Sham Comparator): Participants in the CONTROL group received light touch and BEMER sham treatments. Researchers placed their hands lightly on the subject's cervical paraspinal muscles in the supine position and on the upper thoracic paraspinal muscles in the prone position for approximately 5 minutes. This was done to mimic myofascial release techniques; however, no pressure or action was done. In addition, the subject's laid supine on the BEMER mat (as they would do during a BEMER session), but the device was not activated.
  Interventions: Procedure: Sham OMT + Sham BEMER
- Experimental: Bio Electro-Magnetic Regulation (BEMER) Therapy (Active Comparator): Participants receiving BEMER therapy laid supine on the BEMER mat (BEMER International AG). The BEMER was set at intensity 3 for week 1, intensity 4 for week 2, and intensity 5 for week 3. The B.Pad (BEMER International AG) was placed under their cervical region. B.Pad® settings were set at Program 1 (8 minutes long) in week 1 through week 3. These settings were selected based on the manufacturer's recommendations.
  Interventions: Device: BEMER
- OMT (Osteopathic Manipulative Treatment) (Active Comparator): Participants receiving OMT were treated with a standardized sequence to the areas where somatic dysfunctions were found.
  Interventions: Procedure: OMT
- OMT+BEMER (Experimental): Participants receiving BEMER therapy laid supine on the BEMER mat (BEMER International AG). The BEMER was set at intensity 3 for week 1, intensity 4 for week 2, and intensity 5 for week 3. The B.Pad (BEMER International AG) was placed under their cervical region. B.Pad® settings were set at Program 1 (8 minutes long) in week 1 through week 3. These settings were selected based on the manufacturer's recommendations. OMT was performed prior to BEMER therapy for those in the combined group. Participants were treated with a standardized sequence to the areas where somatic dysfunctions were found.
  Interventions: Device: BEMER; Procedure: OMT

INTERVENTIONS:
Device: BEMER — Bio-Electro-Magnetic Energy Regulation (BEMER) is an emerging therapeutic modality that deploys a biorhythmically defined stimulus through a pulsed electromagnetic field and has been shown to reduce musculoskeletal pain.
  Arms: Experimental: Bio Electro-Magnetic Regulation (BEMER) Therapy; OMT+BEMER
Procedure: OMT — Osteopathic manipulative therapy (OMT) is a form of manual therapy utilized by osteopathic physicians and some allopathic physicians to treat a broad variety of musculoskeletal ailments, including neck pain.
  Arms: OMT (Osteopathic Manipulative Treatment); OMT+BEMER
Procedure: Sham OMT + Sham BEMER — Participants in the CONTROL group received light touch and BEMER sham treatments. Researchers placed their hands lightly on the subject's cervical paraspinal muscles in the supine position and on the upper thoracic paraspinal muscles in the prone position for approximately 5 minutes. This was done to mimic myofascial release techniques; however, no pressure or action was done. In addition, the subject's laid supine on the BEMER mat (as they would do during a BEMER session), but the device was not activated.
  Arms: OMT + BEMER PLACEBO

SUMMARY:
Neck pain is a common ailment in the United States. Although there are several different treatments and approaches to help individuals with neck pain, the number affected by this condition has been steadily increasing.

OMT has been shown to be helpful in the treatment of neck pain. In fact, the use of OMT has been shown to increase mobility of the myofascial tissues, visceral motion and decrease pain in patients with neck pain. Bio Electro-Magnetic Regulation (BEMER) Therapy is a therapeutic modality that deploys a biorhythmically defined stimulus through a Pulsed Electromagnetic Field (PEMF), which leads to an increase in blood flow. The positive effects of BEMER on the circulation has been shown to result in significant increases in arteriovenous oxygen difference, number of open capillaries, arteriolar and venular flow volume, and flow rate of red blood cells in the microvasculature. Therefore, BEMER can potentially be used in the treatment of neck pain by improving microcirculation in muscular tissue. Therefore, it is possible that the combination of OMT and BEMER therapy may provide additive effects in reducing neck pain. The purpose of this study is to investigate the individual and combined effects of OMT and BEMER therapy on neck pain in adults.

DETAILED DESCRIPTION:
Neck Pain is defined as "pain in the neck with or without pain referred to one or both upper limbs that lasts for at least one day". It has been estimated that 66% of the population will suffer from neck pain at some point during their lifetime and has been reported as the fourth leading cause of disability worldwide. There is considerable variation in the reported prevalence rates of neck pain, most likely because of differences in the definition of neck pain and the lack of homogeneity in the studies. Current available studies suggest the one-year estimated incidence of neck pain to range between 10.4% and 21.3%, with a higher incidence noted in computer and office workers. The prevalence of neck pain ranges from 10% to 20%, and the most common cause of neck pain in adults stems from degenerative changes in the cervical spine. Most cases of neck pain tend to run an episodic course over one's lifetime, thus relapses are relatively common.

The differential diagnosis for neck pain is extensive, and a methodical approach is essential to rule out potentially life-threatening conditions. The vast majority of neck pain is not due to organic pathology, and thus, has been termed "non-specific" or "mechanical". Interventions available to manage neck pain include analgesics, physiotherapy, educational modalities, exercise, and manual therapy. While useful in acute, short-term reduction of pain, analgesic therapy such as NSAIDs (nonsteroidal anti-inflammatory drugs) produce significant side effects of gastrointestinal bleeding and cardiovascular events. Use of opioids, while also useful for acute, short-term pain relief, should produce hesitation in prescription due to risk of opioid dependence and hyperalgesia syndromes.

Osteopathic manipulative treatment (OMT) is a fundamental skill set that osteopathic physicians acquire early during their medical training and is widely utilized among practicing osteopathic physicians to treat neck pain and other musculoskeletal complaints. OMT is a unique, hands-on treatment modality used by osteopathic physicians to augment the conventional management of neck pain and has been studied to demonstrate favorable outcomes in the treatment of neck pain.

In addition to conventional treatment modalities, Bio-Electro-Magnetic Energy Regulation (BEMER) therapy (BEMER International AG) has emerged as a proposed therapeutic option. BEMER therapy utilizes a biorhythmically defined stimulus through a pulsed electromagnetic field. BEMER devices operate with unique parameters and are postulated to have a primary effect of improving tissue microcirculation. BEMER therapy leads to an increase in the number of open capillaries, vasomotion of micro vessels, arteriovenous oxygen difference, arteriolar and venular flow volume, and flow rate of red blood cells in a specific microcirculatory area. Multiple studies have demonstrated positive results in musculoskeletal pain management with the utilization of BEMER therapy. One study in particular demonstrated a potential additive, subjective decrease in reported back pain and improved functional ability after treatment with both OMT and BEMER therapy.

The musculoskeletal, lymphatic, and fascial concepts of OMT have long been comprehensively and collectively proposed as the mechanisms by which the therapy provides alleviation of common musculoskeletal ailments. Existing literature suggests benefit from OMT, however, the need for further exploration of manual therapy remains. As previously discussed, BEMER therapy can reduce musculoskeletal pain via enhanced microcirculation. Therefore, it is plausible that the combination of OMT and BEMER therapy may potentially enhance circulation to the vascular beds in myofascial tissue and could substantially reduce neck pain. The objective of this study was to assess the individual and combined effects of OMT and BEMER therapy in patients with non-specific neck pain.

ELIGIBILITY:
Inclusion Criteria:

* LECOM-Bradenton faculty, staff and Students currently enrolled in LECOM- Bradenton's osteopathic medical program, pharmacy program, dental program, and master's program who are currently experiencing neck pain for at least two weeks will be approached for recruitment.

Exclusion Criteria:

* Subjects will be excluded if they have previously participated in the study, are unable to provide informed consent, are currently pregnant, or have a known medical history of any of the following:

  1. Psychiatric conditions
  2. Skin disorders or open wounds precluding skin contact
  3. Fasciitis or fascial tears
  4. Myositis
  5. Neurological symptoms such as numbness, tingling, weakness in upper extremities
  6. Neoplasia
  7. Bone fracture, osteomyelitis, or osteoporosis
  8. Coagulation problem
  9. Deep vein thrombosis
  10. Adrenal diseases/syndromes
  11. Acute upper or lower respiratory infection
  12. Immunosuppressive syndromes
  13. Radiation or chemotherapy within the past 3 years
  14. Lupus
  15. Osteopenia
  16. Congestive heart failure
  17. BMI greater than 30
  18. Any other autoimmune disease not stated above
  19. Medication changes within the last 4 weeks
  20. Asthma exacerbations within the last 4 weeks
  21. Immunosuppressive therapy as a consequence of organ transplantation
  22. Immunosuppressive therapy as a consequence of allogeneic cellular transplantations or bone marrow stem cell transplantation
  23. Other conditions often requiring immunosuppressive therapy
  24. Anticoagulant therapy
  25. Known sensitivity to the carotid sinus reflex
  26. Advanced carotid disease
  27. Down syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Lorenzo, PhD, MS, Principal Investigator — Lake Erie College of Osteopathic Medicine
Locations (1):
- Lake Erie College of Osteopathic Medicine, Bradenton, Florida, United States

REFERENCES:
- [Derived] Palmer GM, Dominick N, Kane M, Bawek S, Burch B, Sanders T, Phrathep D, Myers N, Lorenzo S. Effect of osteopathic manipulative treatment and Bio-Electro-Magnetic Energy Regulation (BEMER) therapy on generalized musculoskeletal neck pain in adults. J Osteopath Med. 2023 Dec 1;124(4):153-161. doi: 10.1515/jom-2023-0128. eCollection 2024 Apr 1. PMID 38033194

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OMT + BEMER PLACEBO | Experimental: Bio Electro-Magnetic Regulation (BEMER) Therapy | OMT (Osteopathic Manipulative Treatment) | OMT+BEMER
Started | 12 | 12 | 10 | 10
Completed | 8 | 10 | 10 | 10
Not Completed | 4 | 2 | 0 | 0
Not completed — error in completing survey | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OMT + BEMER PLACEBO | Experimental: Bio Electro-Magnetic Regulation (BEMER) Therapy | OMT (Osteopathic Manipulative Treatment) | OMT+BEMER | Total
Number analyzed (Participants) | 12 | 12 | 10 | 10 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 10 | 10 | 44
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (1.6) | 24.6 (1.6) | 25.9 (2.5) | 24.8 (1.8) | 25.2 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 7 | 8 | 32
  Male | 4 | 3 | 3 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 12 | 12 | 10 | 10 | 44
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 10 | 10 | 44
Visual Analog Scale [Mean (Standard Deviation); unit: units on a scale] — Scale range (0-100) to determine level of pain (0:no pain, 100: the most pain ever experienced)
  units on a scale | 20.3 (20.2) | 13.2 (14.0) | 16.5 (13.8) | 32.9 (33.4) | 20.7 (20.4)

OUTCOME MEASURES:

1. Primary Outcome: Neck Pain Rating Neck Disability Index (NDI)
Description: Assessed by questionnaire rating, compared with pre-intervention rating Neck Disability Index (NDI). Score ranges 0-50. Minimum score=0 (no activity limitation), Maximum score=50 (complete activity limitation). Lower scores is better as it reflect lower activity limitation
Time Frame: Within 1 week of completion of 3-week intervention period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMT + BEMER PLACEBO | Experimental: Bio Electro-Magnetic Regulation (BEMER) Therapy | OMT (Osteopathic Manipulative Treatment) | OMT+BEMER
Number analyzed (Participants) | 8 | 10 | 10 | 10
units on a scale | 13 (7.6) | 7.4 (8.5) | 12.2 (10.9) | 11.2 (7.6)

2. Primary Outcome: Neck Pain Rating Visual Analog Scale (VAS)
Description: Assessed by questionnaire rating, compared with pre-intervention rating Visual Analog Scale (VAS). Score ranges 0-100. Minimum score=0 (no pain), Maximum score=100 (worst pain ever felt). Lower scores is better as it reflect lower pain
Time Frame: Within 1 week of completion of 3-week intervention period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMT + BEMER PLACEBO | Experimental: Bio Electro-Magnetic Regulation (BEMER) Therapy | OMT (Osteopathic Manipulative Treatment) | OMT+BEMER
Number analyzed (Participants) | 8 | 10 | 10 | 10
units on a scale | 15.5 (13.4) | 7.1 (10.8) | 16 (14.2) | 11.5 (8.4)

3. Primary Outcome: Quality of Life Rating Short Form 12-item (SF-12) Health Survey
Description: Assessed by questionnaire rating, compared with pre-intervention rating Short form 12-item (SF-12) health survey. Scores range 0%-100%. Score of 0 (minimum) no pain. Score of 100 (maximum) lot of pain. Lower scores is better as it reflect lower pain
Time Frame: Within 1 week of completion of 3-week intervention period
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMT + BEMER PLACEBO | Experimental: Bio Electro-Magnetic Regulation (BEMER) Therapy | OMT (Osteopathic Manipulative Treatment) | OMT+BEMER
Number analyzed (Participants) | 8 | 10 | 10 | 10
units on a scale | 47.5 (11.1) | 45.4 (9) | 43.7 (14.7) | 45.6 (13)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | OMT + BEMER PLACEBO | Experimental: Bio Electro-Magnetic Regulation (BEMER) Therapy | OMT (Osteopathic Manipulative Treatment) | OMT+BEMER
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/39/NCT05889039/Prot_SAP_ICF_001.pdf